CLINICAL TRIAL: NCT06051474
Title: Treating Nicotine Addiction in Caregivers of Children at American Family Children's Hospital
Brief Title: Treating Caregivers Who Smoke at AFCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0727; SMPH\PEDIATRICS\PED HOSP (Other: UW Madison); Protocol Version 5/23/23 (Other: UW Madison)
Record Dates: First submitted 2023-09-12; First posted 2023-09-25 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Smoking; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Caregivers of hospitalized children (Experimental)
  Interventions: Drug: Nicotine Replacement Product

INTERVENTIONS:
Drug: Nicotine Replacement Product — Adults will receive a 2-week supply of nicotine patches to place on skin (14mg or 21mg; dosing depending on tobacco use per package insert) and oral nicotine mini-lozenges (2mg, 4mg, dosing depending on tobacco use per package insert). All participants will also receive a single smoking cessation counseling session with a physician. Surveys will be completed pre-intervention, within 24 hours of hospital discharge, and 2-weeks after hospital discharge.

SUMMARY:
The purpose of this research study is to 1) see if a smoking cessation program is something that caregivers will use while their child is hospitalized, 2) see if caregivers think this program is something we should institute across the hospital, and 3) see if this program can help caregivers reduce their smoking.

Participants will:

* Complete a survey regarding smoking behavior and thoughts about quitting;
* Undergo a 20-minute counseling session; and,
* Use nicotine patches and mini-lozenges for 2 weeks

DETAILED DESCRIPTION:
All participants will receive a one-time visit with the study physician. This visit will consist of a brief counseling session. Counseling sessions will last approximately 20 minutes and cover the 3 objectives of 1) review participants' motivation for smoking and for quitting; 2) use the information on participants' motives to provide tailored education regarding a) benefits of quitting smoking to the caregiver and the child, b) strategies to reduce nicotine withdrawal symptoms/urges to smoke during the hospitalization, and c) benefits of smoke-free home and car rules; and, 3) review smoking cessation resources.

After the counseling session, participants will be provided a 2-week supply of nicotine patches and nicotine mini-lozenges, along with instructions for their use. The study physician will review how to use the medication, dosing, benefits of use, and potential side effects of use.

Within 24 hours of discharge, participants will be contacted to complete a post-intervention survey, which will assess nicotine replacement therapy (NRT) use during the hospitalization and likelihood that the participant would recommend program implementation in the hospital. Smoking behavior during the child's hospitalization will be examined, including assessments of 1) number of cigarettes smoked per day and 2) number of times participant left the child's bedside to smoke per day. Participant's self-efficacy and interest in quitting smoking will be assessed, using the same questions from the pre-intervention survey, to assess for changes after the intervention.

Participants will be contacted 2 weeks after discharge with a link to complete the follow-up survey to again assess current smoking status, use of NRT post-hospitalization, self-efficacy and interest in quitting smoking, establishment of smoke-free home and car rules, and interest in ongoing smoking cessation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized child will have a 'yes' response to the screening question, "Does anyone in your household smoke"
* Hospitalized child is expected to be admitted for >24 hours
* Caregiver is at least 18 years of age
* Participant self-identifies as the primary caregiver of the hospitalized child during the hospitalization
* Participant smokes ≥5 cigarettes per day
* Participant is willing and able to use NRT
* Participant is not currently pregnant, trying to get pregnant, or breastfeeding and willing to use acceptable birth control for duration of medication use
* Participant is willing to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

* Contraindication to NRT use (pregnancy, myocardial infarction in past 2 weeks)
* Previous reaction to the nicotine patch or mini-lozenge that prevented them from continuing to use it
* Current use of smoking cessation medications (any NRT, bupropion, varenicline)
* Caregiver's child is being cared for by study physician (Dr. Brian Williams)
* Need for an interpreter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Enrollment in study | Study recruitment, approximately 6 months
  Enrollment will be measured as a relation between the number of people invited to enroll versus the number who enroll
NRT use | 2 weeks post-discharge
  Number of participants who use the NRT provided
Acceptability of smoking intervention | 2 weeks post-discharge
  Self-report by participant via survey. Score ranges from 1-7, with 1 indicating would not recommend implementing cessation program and 7 indicating definitely recommend implementing program.

SECONDARY OUTCOMES:
Change in number of cigarettes smoked per day | Baseline to 2 weeks post-discharge
  Self-report by participants via survey
Number of times participant left child's bedside to smoke | From admission to discharge, up to 4 weeks
  Self-report by participant via survey
Change in self-confidence in quitting smoking | Baseline to 2 weeks post-discharge
  Self-report by participant via survey. Score ranges from 1-7, with 1 indicating no confidence in ability to quit smoking and 7 indicating extreme confidence.
Change in motivation to quit smoking | Baseline to 2 weeks post-discharge
  Self-report by participant via survey. Score ranges from 1-7, with 1 indicating no motivation to quit smoking and 7 indicating extreme motivation.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Williams, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- American Family Children's Hospital, Madison, Wisconsin, United States